CLINICAL TRIAL: NCT01205256
Title: IRB-HSR# 14145 R,S Methadone: Analgesia and Pharmacokinetics in Adolescents Undergoing Scoliosis Correction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Christopher Stemland, MD, Attending Anesthesiologist, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 14145
Record Dates: First submitted 2010-09-16; First posted 2010-09-20 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Scoliosis
Keywords: Methadone pharmacokinetics in adolescents
MeSH Terms: conditions — Scoliosis | interventions — Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Methadone (Experimental): 0.25mg/kg IV of racemic methadone at the induction of anesthesia.
  Interventions: Drug: methadone

INTERVENTIONS:
Drug: methadone — 0.25mg/kg IV of racemic methadone at the induction of anesthesia.
  Other Names: 0.25mg/kg IV of racemic methadone

SUMMARY:
This is a pilot study to determine the pharmacokinetics of (R,S) methadone in adolescents. A total of approximately 15 patients will be required. The purpose is to determine the levels of R, S methadone at various time intervals after drug administration. Patients will receive methadone 0.25 mg/kg IV at induction and a standardized anesthetic of remifentanil and propofol. At the conclusion of surgery (45 minutes prior to the completion), the patients will receive a loading dose of morphine based on respiratory rate. A morphine PCA will be utilized for postoperative analgesia. Pharmacokinetic data will be collected in addition to VAS scores, patient and parental satisfaction with analgesia, and a functional pain assessment.

DETAILED DESCRIPTION:
Study Procedures Following Surgery:

* VAS scores will be recorded at intervals of 1,2,3,4,5,6,8,12,16,20,24, 36, 48 , 72 hrs (after extubation).
* Blood samples for PK will require 5ml per sample and may be obtained from an existing IV or direct phlebotomy and will be obtained at 0min, 5min, 10 min, 15min, 20 min, 40 min, 1hr, 2hrs, 3hrs, 4hrs, 5hrs, 6hrs, 8hrs, 10 hrs, 12hrs, 24hrs, 48 hrs, 72hrs, and 96hrs after study drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric scoliosis surgery secondary idiopathic scoliosis, congenital scoliosis,
* Age 12 - 19 inclusive
* ASA class I-II.

Exclusion Criteria:

* Preoperative opioid therapy in previous 2 weeks
* Known hepatic or renal impairment
* Inability to assess pain score due to neurological impairment, hearing impairment
* Allergy to methadone, morphine, fentanyl, propofol or remifentanil
* Pregnant or nursing
* Taking SSRI's, MAOI,anticonvulsants, gabapentin or lyrica
* ASA III or greater patients are excluded
* pre-existing chronic pain

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2009-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
methadone levels | 0min, 5min, 10 min, 15min, 20 min, 40 min, 1, 2hrs, 3hrs, 4hrs, 5hrs, 6hrs, 8hrs, 10 hrs, 12hrs, 24hrs, 48 hrs, 72hrs, and 96hrs.
  Tmax (time to maximum methadone concentration) Cmax (maximum concentration) T1/2 (half-life) AUC last (area under the curve from time 0 to last sample point) AUC inf (area under the curve from time 0 to infinity) VZ (Volume of distribution in the terminal phase) CL (clearance)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Stemland, MD, Principal Investigator — UVA Anesthesiology
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gourlay GK, Willis RJ, Wilson PR. Postoperative pain control with methadone: influence of supplementary methadone doses and blood concentration--response relationships. Anesthesiology. 1984 Jul;61(1):19-26. PMID 6742480
- [Background] Gourlay GK, Wilson PR, Glynn CJ. Pharmacodynamics and pharmacokinetics of methadone during the perioperative period. Anesthesiology. 1982 Dec;57(6):458-67. doi: 10.1097/00000542-198212000-00005. No abstract available. PMID 6128949
- [Background] Claar RL, Walker LS. Functional assessment of pediatric pain patients: psychometric properties of the functional disability inventory. Pain. 2006 Mar;121(1-2):77-84. doi: 10.1016/j.pain.2005.12.002. Epub 2006 Feb 9. PMID 16480823
- [Background] Walker LS, Greene JW. The functional disability inventory: measuring a neglected dimension of child health status. J Pediatr Psychol. 1991 Feb;16(1):39-58. doi: 10.1093/jpepsy/16.1.39. PMID 1826329
- [Background] Vinik HR, Kissin I. Rapid development of tolerance to analgesia during remifentanil infusion in humans. Anesth Analg. 1998 Jun;86(6):1307-11. doi: 10.1097/00000539-199806000-00033. PMID 9620525
- [Background] Davis AM, Inturrisi CE. d-Methadone blocks morphine tolerance and N-methyl-D-aspartate-induced hyperalgesia. J Pharmacol Exp Ther. 1999 May;289(2):1048-53. PMID 10215686
- [Background] Holtman JR Jr, Wala EP. Characterization of the antinociceptive and pronociceptive effects of methadone in rats. Anesthesiology. 2007 Mar;106(3):563-71. doi: 10.1097/00000542-200703000-00022. PMID 17325516
- [Background] Berde CB, Beyer JE, Bournaki MC, Levin CR, Sethna NF. Comparison of morphine and methadone for prevention of postoperative pain in 3- to 7-year-old children. J Pediatr. 1991 Jul;119(1 Pt 1):136-41. doi: 10.1016/s0022-3476(05)81054-6. PMID 2066846
- [Background] Shir Y, Shenkman Z, Shavelson V, Davidson EM, Rosen G. Oral methadone for the treatment of severe pain in hospitalized children: a report of five cases. Clin J Pain. 1998 Dec;14(4):350-3. doi: 10.1097/00002508-199812000-00013. PMID 9874015
- [Background] Dale O, Hoffer C, Sheffels P, Kharasch ED. Disposition of nasal, intravenous, and oral methadone in healthy volunteers. Clin Pharmacol Ther. 2002 Nov;72(5):536-45. doi: 10.1067/mcp.2002.128386. PMID 12426517